CLINICAL TRIAL: NCT03882242
Title: Impact on Self-esteem, Body Image and Media Literacy of Facilitators in the Program "In Favor of Myself" - Quantitative and Qualitative Longitudinal Research
Brief Title: Effect of a Prevention Program on Program Facilitators
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: telhai
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Self Esteem; Body Image

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Program Facilitators (Experimental): Participants will learn about and deliver (facilitate) a prevention program "In favor of Myself" to school-children
  Interventions: Behavioral: Facilitation of a school-based program

INTERVENTIONS:
Behavioral: Facilitation of a school-based program — Participants deliver the prevention program (described in previous research) to school-children.

SUMMARY:
The study will examine, through quantitative and qualitative research, how the delivery of the program "In Favor of Myself" to school children influences the program facilitators themselves, and the effect on their self-esteem, body-image, and media literacy.

DETAILED DESCRIPTION:
In recent decades, the existence of prevention and intervention programs has gained momentum and has become an important part of our culture. Programs are delivered around the world in a wide variety of fields and subjects. They serve as an auxiliary tool for the improvement, awareness, empowerment, treatment and response to a range of social and personal behavioral issues and behaviors, eradication of harmful behaviors, and more.

In the literature there is ample evidence and proof of the nature of the effects and impact of different programs on the group of participants involved. Many successes in these programs relate to the contents of the program, the level of interest among the participants, the way the program is delivered, the degree of interaction between the facilitators and the participants, and more.

Yet there is little reference in the literature to the aspect that examines the program facilitators themselves and the potential impact that the programs will have on a variety of aspects and personal measures in the lives of the facilitators. Among these measures is the experience of instruction, including the experience of teaching and learning embodied in it, the involvement of the ego and the involvement of the facilitator in the tasks, the impact on the values and the personal level of the facilitators, including impact on their self-esteem.

This study will examine, through quantitative and qualitative research, how the delivery of the program "In Favor of Myself" to school children influences the program facilitators themselves, and the effect on their self-esteem, body-image, and media literacy.

The research hypothesis is that the self-esteem, body image, media literacy, the sense of ability, and personal empowerment of the group of facilitators who delivered the program will be increased, and their behavior will change according to the subjects of the program.

ELIGIBILITY:
Inclusion Criteria:

* College students participating in the relevant course
* Completed study questionnaire before and after delivering the prevention program.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Rosenberg Self Esteem Scale (RSE) | Measured twice over three months: Before beginning of program and after program ends.
  Rosenberg Self Esteem Scale (Rosenberg, 1965)- 10 items. Scoring involves a method of combined ratings. Low self-esteem responses are "disagree" or
  "strongly disagree" on items 1, 3, 4, 7, 10, and "strongly agree" or "agree" on items 2, 5, 6, 8, 9. Two or three out of three correct responses to items 3, 7, and 9 are scored as one item. One or two out of two correct responses for items 4 and 5 are considered as a single item; items 1,8, and 10 are scored as individual items; and combined correct responses (one or two out of two) to items 2 and 6 are considered to be a single item.
Change from Baseline in Contingencies of Self Worth Scale (CSW) | Measured twice over three months: Before beginning of program and after program ends.
  Contingencies of Self Worth Scale- 25 items (Crocker et al., 2003). We used 2 subscales: Appearance and Approval from others.
Change from Baseline in Sociocultural Attitudes Towards Appearance Questionnaire-3 (SATAQ-3) | Measured twice over three months: Before beginning of program and after program ends.
  The Sociocultural Attitudes Towards Appearance Questionnaire (Schaefer et al., 2015). The investigators included 3 subscales: Internalization - Thin/Low Body Fat, Internalization - Muscular/Athletic, Pressures - Media- 14 items. Items are rated on a 5-point scale: (1) always, (2) often, (3) sometimes, (4) rarely, (5) never. The total score is based on computing the average. A higher score indicates higher pressure from the media to change one's look.
Change from Baseline in Advertising Scale | Measured twice over three months: Before beginning of program and after program ends.
  The Advertising scale contains 1 item- Identification of strategies used by media. This question is reflected as a protective factor. It contains 8 different strategies which participants choose from: higher number of strategies identified indicate better media literacy. (Golan et al., 2013).
Change from Baseline in Eating Disorders Inventory 2- Drive for Thinness | Measured twice over three months: Before beginning of program and after program ends.
  The EDI-2 Drive for Thinness sub-scale which includes 7 items. The items are rated on a 6-point scale: (1) never, (2) rarely, (3) sometimes, (4) often, (5) usually, and (6) always.The final score is computed by summing the points. Higher scores indicate a higher drive for thinness.
Change from Baseline in Eating Attitudes Test | Measured twice over three months: Before beginning of program and after program ends.
  Eating Attitudes Test- 26 items The Eating Attitudes validated scale for children and adolescents. The items are rated on a 6-point scale: (1) never, (2) rarely, (3) sometimes, (4) often, (5) usually, and (6) always. Scores above 20 indicates a high level of concern about dieting, body weight, or problematic eating behaviors. (Maloney, McGuire, & Daniels, 1988)
Change from Baseline in Body Esteem Scale | Measured twice over three months: Before beginning of program and after program ends.
  Body Esteem Scale- This questionnaire examines self-esteem of body and physical appearance and consists of 3 subscales: appearance (10 items), weight (8 items) and attribution 187 to others (5 items). Items are rated on a 5-point scale: (1) never, (2) rarely, (3) sometimes, (4) 188 often, and (5) always. A higher score indicates higher body-esteem (Mendelson, Mendelson, & White, 2001)
Semi-structured interviews | Measured once for 90 minutes, after completion of program delivery.
  A qualitative semi-structured interview is to be performed with 10 facilitators after delivery of the program. The interview will be conducted by a research student following guided instructions. The duration of the personal interview will be 90 minutes, will be recorded, completed and analyzed according to the qualitative research rules.